CLINICAL TRIAL: NCT04834453
Title: Correlation of Trans Cranial Doppler Ultrasound and CT Scan in Monitoring of Posttraumatic Brain Edema
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant professor, Ain Shams University
Other Study IDs: R 75/2021
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Brain Edema
MeSH Terms: conditions — Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transcranial ultrasound — - Transcranial Doppler sonography will be performed with the patients in the supine position., using low frequency probe of 2 MHz will be placed on temporal bone- will be performed daily

SUMMARY:
The most common tool for diagnosis and follow up of cerebral edema in ICU is brain CT scan that necessitate patient transportation with risk of hemodynamic instability, and exposure to radiation.

Transcranial Doppler (TCD) sonography allows true and rapid imaging of blood flow velocities of intracranial vessels. Transcranial Doppler sonography provides noninvasive evaluation of intracranial pressure by its characteristic wave patterns

ELIGIBILITY:
Inclusion Criteria:

* isolated blunt Traumatic Brain Injury
* age 18-60 years

Exclusion Criteria:

* Pregnancy
* Intracerebral hemorrhage
* Patients whose blood flow velocities could not be obtained from Trans temporal acoustic bone windows.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with isolated blunt TBI from (age 18-60 years) of both sex, will be included in the study and followed prospectively. Severity of trauma is evaluated by GCS, Rotterdam computed tomography score (CTS) care system with the help of our radiodiagnosis colleagues
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
the correlation between CCT scans score and Pulsatility Index of each patient | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] Ammar MA, Abdelmoneim W, Abdalla W. Correlation of transcranial Doppler based parameters with computed tomography assessed cerebral oedema score in patients with traumatic brain injury: A prospective observational study. Indian J Anaesth. 2023 Feb;67(2):180-185. doi: 10.4103/ija.ija_337_22. Epub 2023 Feb 16. PMID 37091450